CLINICAL TRIAL: NCT01783691
Title: A Single Ascending Dose Phase 1 Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Biologic Activity of Intravenous NKTT120 in Adults With Stable Sickle Cell Disease
Brief Title: Safety, Pharmacokinetic, and Pharmacodynamic Study of NKTT120 in Adult Patients With Stable Sickle Cell Disease (SCD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NKT Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120-SCD1
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — NKTT120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NKTT120 (Experimental)
  Interventions: Drug: NKTT120

INTERVENTIONS:
Drug: NKTT120

SUMMARY:
The purpose of this study is to determine the safety, pharmacokinetics, and pharmacodynamics of NKTT120 in adult patients with stable sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Subject has a confirmed diagnosis of HbSS or HbSβ0thal
* Subject has stable SCD defined as not having acute VOC, ACS, or other major SCD associated event during the month prior to enrollment

Exclusion Criteria:

* Subject had an SCD-related VOC or ACS that required hospitalization or treatment in acute care outpatient setting in the month prior to enrollment
* Subject requires a program of prescheduled regularly administered packed red blood cell (pRBC) transfusions or Subject received a pRBC transfusion in the month prior to enrollment
* Subject has evidence of latent or active tuberculosis
* Subject has a major concurrent illness or medical condition
* Subject is pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by (1) adverse events (2) laboratory values (3) vital signs and (4) physical exam. | 180 days

SECONDARY OUTCOMES:
Pharmacokinetics assessed by plasma drug concentration levels | 0; 15, 30, 60 minutes; 3,6, hours; 1,2,3,7,14,30,60,90 days
Pharmacodynamics as measured by assessments of peripheral blood lymphocyte subsets | 0, 0.25, 1, 2, 7, 14, 30, 60, 90, 120 days

OTHER OUTCOMES:
Pain scores as assessed by daily electronic diary | Daily for 120 days
Quality of Life as assessed by two separate Quality of Life instruments | 0, 30, 60, 90, 120 days
Lung function as measured by pulmonary function tests | 0; 30 minutes; 30, 60, 90, 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Mazanet, MD, Study Director — NKT Therapeutics
Locations (6):
- United States (6):
  - Children's Hospital & Research Center at Oakland, Oakland, California
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - UNC Sickle Cell Program, Chapel Hill, North Carolina
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Field JJ, Majerus E, Ataga KI, Vichinsky EP, Schaub R, Mashal R, Nathan DG. NNKTT120, an anti-iNKT cell monoclonal antibody, produces rapid and sustained iNKT cell depletion in adults with sickle cell disease. PLoS One. 2017 Feb 2;12(2):e0171067. doi: 10.1371/journal.pone.0171067. eCollection 2017. PMID 28152086